CLINICAL TRIAL: NCT02210754
Title: Characterization of Nicotine Exposure and Urge-to-Smoke Following a Single Controlled Administration and Short-Term Ad Lib Use of Electronic Cigarettes and Conventional Cigarettes in Adult Smokers
Brief Title: Characterization of Nicotine Exposure and Urge-to-Smoke Following Use of Electronic and Conventional Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lorillard Tobacco Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: Galileo
Record Dates: First submitted 2014-07-30; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Smoking
Keywords: Nicotine; Pharmacokinetics; Pharmacodynamics; blu e-cigs; Tolerability; Safety; Smoke urge
MeSH Terms: conditions — Smoking | interventions — Nicotine; Glycerol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- E-cigarette 1 (Experimental): blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin vehicle)
  Interventions: Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/PG vehicle); Other: Marlboro Cigarette
- E-cigarette 2 (Experimental): blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/propylene glycol (PG) vehicle)
  Interventions: Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin vehicle); Other: blu™ Magnificent Menthol rechargeable (2.4% nicotine, glycerin vehicle); Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin/PG vehicle); Other: Marlboro Cigarette
- E-cigarette 3 (Experimental): blu™ Magnificent Menthol rechargeable (2.4% nicotine, glycerin vehicle)
  Interventions: Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/PG vehicle); Other: Marlboro Cigarette
- E-cigarette 4 (Experimental): blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin vehicle)
  Interventions: Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin/PG vehicle); Other: Marlboro Cigarette
- E-cigarette 5 (Experimental): blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin/PG vehicle)
  Interventions: Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/PG vehicle); Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin vehicle); Other: Marlboro Cigarette
- Combustible Cigarette (Active Comparator): Marlboro Cigarette
  Interventions: Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin vehicle); Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/PG vehicle); Other: blu™ Magnificent Menthol rechargeable (2.4% nicotine, glycerin vehicle); Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin vehicle); Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin/PG vehicle)

INTERVENTIONS:
Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin vehicle) — electronic cigarettes
  Arms: Combustible Cigarette; E-cigarette 2
Other: blu™ Classic Tobacco rechargeable (2.4% nicotine, glycerin/PG vehicle) — electronic cigarettes
  Arms: Combustible Cigarette; E-cigarette 1; E-cigarette 3; E-cigarette 5
Other: blu™ Magnificent Menthol rechargeable (2.4% nicotine, glycerin vehicle) — electronic cigarettes
  Arms: Combustible Cigarette; E-cigarette 2
Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin vehicle) — electronic cigarettes
  Arms: Combustible Cigarette; E-cigarette 5
Other: blu™ Classic Tobacco rechargeable (1.6% nicotine, glycerin/PG vehicle) — electronic cigarettes
  Arms: Combustible Cigarette; E-cigarette 2; E-cigarette 4
Other: Marlboro Cigarette — cigarettes
  Arms: E-cigarette 1; E-cigarette 2; E-cigarette 3; E-cigarette 4; E-cigarette 5

SUMMARY:
This trial was the initial characterization of the blu™ products being studied, with the purpose of gaining an understanding of the exposure to nicotine and craving reduction attained following use of blu™ e-cigarettes by adult smokers. Two types of exposures were utilized: a single controlled administration and a short-term ad lib use. As smoking behaviors vary from smoker to smoker, a controlled administration allows for some standardization of nicotine "dose" for each of the study products to better understand their uptake characteristics as well as urge reduction achieved under controlled conditions. Further evaluation under ad lib product use conditions provides insight into product self-administration behaviors that will allow subjects to achieve acceptable levels of urge reduction. Comparisons were made to evaluate differences between blu™ formulations as well as to the market-leading conventional cigarette, Marlboro Gold King Size ("Marlboro cigarette').

DETAILED DESCRIPTION:
This was a randomized, partially single-blinded, 6-period crossover study of 24 subjects.

The primary objectives of this study were to:

1. characterize the rate and extent of nicotine exposure following a single controlled administration and ad lib use of blu™ e-cigarettes,
2. characterize smoking urge following a single controlled administration and ad lib use of blu™ e cigarettes.

The secondary objectives of this study were to:

1. Compare the pharmacokinetic (PK) profile of nicotine between selected blu™ formulations and between the blu™ products and Marlboro cigarettes following a single controlled administration and ad lib use of each study product.
2. Compare changes in smoking urge within and between selected blu™ formulations and between the blu™ products and Marlboro cigarettes following a single controlled administration and ad lib use of each study product.
3. Compare the changes in exhaled carbon monoxide (CO) within and between selected blu™ formulations and between the blu™ products and Marlboro cigarettes following use of each study product.
4. Assess the tolerability of each study product following short-term use.

Subjects were provided blu™ Classic Tobacco and Magnificent Menthol products containing 2.4% nicotine, glycerin vehicle for 1 week prior to participation in the study to familiarize themselves with the use of the products. Subjects were confined to the clinic for the entire study duration and abstained from use of nicotine containing products for a period of at least 36 hours prior to each product administration. Each product administration included a controlled product administration and a 1 hour ad lib use of the study products. The controlled product administration consisted of 50 inhalations of the assigned e-cigarette product (5-second inhalations at 30-second intervals) or smoking one Marlboro cigarette (30-second intervals with the subjects' normal inhalation duration) with inhalations monitored by the clinical staff. The start of the ad lib product use was 30 minutes following the start of the controlled product use. During ad lib use, subjects were allowed to self-administer the e-cigarette product as desired for the entire hour and were responsible for maintaining their own inhalation counts. During the ad lib cigarette product use, subjects requested the product from the staff as desired and maintained their own inhalation counts.

Pharmacokinetics: Blood samples for the measurement of plasma nicotine concentrations were taken by direct venipuncture at 10 minutes prior to, and 5, 10, 15, 20, 25, 30, 45, 60, 75, and 90 minutes following the start of the controlled product administration. Non-compartmental PK parameters such as Peak Plasma Concentration and Area under the Plasma Concentration versus time curve were calculated from the plasma nicotine concentration-time data.

Pharmacodynamics: Smoking urge was assessed using a 100 mm visual analog scale (VAS). Assessments occurred within 1 minute prior to the -10 (pre-product administration), 5, 15, 25, 30, 60, and 90-minute PK blood draws. The following non-compartmental Pharmacodynamic parameters were calculated from the smoking urge change-from-baseline data: Emax0-30, Emaxreduction0-30, AUEC0-30, tEmax0-30, AUEC30-90, and E90.

Other Measurements: Exhaled CO measurements occurred at approximately 20 minutes prior to the start of the controlled product use and at approximately 15 minutes following the end of the ad lib product use.

Tolerability: Adverse events, physical examinations, vital signs, ECGs, and laboratory safety tests were assessed to evaluate enrolment criteria and subject safety during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female smokers
* 21 to 65 years of age, inclusive, at Screening.
* Smoker for at least 12 months prior to Check-in
* Currently smoked an average of 10 or more manufactured cigarettes per day (no restriction on brand-style, king size [ approx. 83 - 85 mm] and 100s [approximately 98 - 100 mm] only)
* A history of e-cigarette use was allowed.
* Females of childbearing potential agreed to use a PI-approved method of contraception

Exclusion Criteria:

* Use of tobacco- or nicotine-containing products other than manufactured cigarettes and e-cigarettes (e.g., roll-your-own cigarettes, bidis, snuff, snus, tablets, inhalers, pipes, cigars, chewing tobacco, nicotine replacement therapies [e.g., gum, patches, lozenges, nasal spray, or inhalers]) within 28 days prior to Day 1 product administration or during the study.
* Use of any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or buproprion (Zyban®) within 3 months prior to Day 1 product administration and throughout the study.
* Known hypersensitivity to menthol, glycerol, or propylene glycol (PG).
* Exhaled CO ≤ 10 ppm at Screening.
* Self-reported puffers (i.e., smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
* Use of medications known to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, desipramine, isoniazid, ketoconazole, miconazole, phenobarbital, rifampin, tranylcypromine, and methoxsalen) within 3 months prior to Day 1 product administration.
* History of drug or alcohol abuse within 24 months of Day 1 product administration
* Female subjects who were pregnant, lactating, or intended to become pregnant from Screening through completion of study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Profile nicotine pharmacokinetics following use of e-cigs and regular cigarettes | 6 months
  Measure plasma nicotine PK outcome measures such as Peak Plasma Concentration and Area under the Plasma Concentration versus time curve.

SECONDARY OUTCOMES:
Assess smoking urge scores on the Visual Analog Scale following use of electronic and regular cigarettes | 6 months
  Smoking urge was assessed using a 100 mm visual analog scale (VAS). Assessments occurred within 1 minute prior to the -10 (pre-product administration), 5, 15, 25, 30, 60, and 90-minute PK blood draws on Days 1, 3, 5, 7, 9, and 11. The 30-minute assessment was intended to coincide with the start of the ad lib product use. The following non-compartmental pharmacodynamic parameters were calculated from the smoking urge change-from-baseline data: Maximum smoking urge reduction and change-from-baseline from time zero to 30 minutes, area under the effect curve (smoking urge change-from-baseline) from time 0 to 30 minutes and 30 to 90 minutes,time of the maximum (positive or negative) smoking urge change-from-baseline from time 0 to 30 minutes and Observed smoking urge change-from-baseline at 90 minutes.

OTHER OUTCOMES:
Evaluation of the Number of Participants with Adverse Effects, Vital Signs, and Concomitant Medications | 6 months
  AE seriousness, severity, and relationship to study product were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Gartner, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] D'Ruiz CD, Graff DW, Yan XS. Nicotine delivery, tolerability and reduction of smoking urge in smokers following short-term use of one brand of electronic cigarettes. BMC Public Health. 2015 Sep 30;15:991. doi: 10.1186/s12889-015-2349-2. PMID 26424091